CLINICAL TRIAL: NCT04060836
Title: Randomized, Open-label, Double Cycle, Crossover, Pharmacokinetics Study of Recombinant Coagulation Factor VIII Injection Versus Xyntha® in Subjects With Hemophilia A.
Brief Title: Pharmacokinetics Evaluation of Recombinant Coagulation Factor VIII Injection in Subjects With Hemophilia A.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CTTQ-NXBYZ-02-PK
Record Dates: First submitted 2019-07-16; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Participants will be assigned to group A or B with a scale of 1:1 , i.e. infuse reference drug Xyntha (group A), then experimental drug (group B). All participants who completed the study will enter the prophylaxis group study.
  Interventions: Drug: Xyntha; Drug: Recombinant Coagulation Factor VIII Injection
- group B (Experimental): Participants will be assigned to group A or B with a scale of 1:1 , i.e. infuse experimental drug (group B), then reference drug Xyntha (group A). All participants who completed the study will enter the prophylaxis group study.
  Interventions: Drug: Xyntha; Drug: Recombinant Coagulation Factor VIII Injection

INTERVENTIONS:
Drug: Xyntha — Recombinant Coagulation Factor VIII Injection produced by Pfizer Inc.
Drug: Recombinant Coagulation Factor VIII Injection — A kind of Recombinant Coagulation Factor VIII Injection produced by sponsor.

SUMMARY:
This is a multi-center, open-label, randomized study. Participants will be assigned to A or B groups with a scale of 1:1 , i.e. infuse study drug followed by Xyntha (group A), or the alternate sequence (group B). All participants who completed the study will enter the Prophylactic Therapy Study.

ELIGIBILITY:
Inclusion Criteria:

1. Hemophilia A.
2. FVIII:C <1%. 3）12 and 65 years old.

4）Has received FVIII treatment and the treatment exposure days ≥100. 5）Has bleeding treatment records of at least 3 months before randomization. 6）FVIII inhibitor assay results is negative.

7） Subjects should agree to use an adequate method of contraception during the study.

8）Understood and Signed an informed consent form. 9）Has not received an treatment of any FVIII within 4 days before the first dose.

10）Non-bleeding state.

Exclusion Criteria:

1. Has a history or family history of blood coagulation factor VIII inhibitor.
2. Has other coagulation dysfunction diseases in addition to hemophilia A.
3. HIV positive.
4. Plan to receive surgery during the trial.
5. Has used immunomodulator within one weeks before the first dose，and less than 7 half-life periods.
6. Known to be allergic to experimental drugs or any excipients.
7. Severe anemia and need blood transfusion.
8. Serious liver or kidney damage.
9. Serious heart disease.
10. Uncontrollable hypertension.
11. Has participated in other clinical studies within one month before the first dose.
12. The researchers believe that it is not suitable for participants.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters between test preparation and reference preparation, peak plasma concentration (Cmax) | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on single dose in day 1 to day 4.
  Cmax is the maximum plasma concentration of Recombinant Coagulation Factor VIII or metabolite(s).
Pharmacokinetic parameters between Recombinant Coagulation Factor VIII, Area under the plasma concentration verus time curve(AUC) | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on single dose in day 1 to day 4.
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of area under the plasma concentration time curve from zero to infinity.
Incremental recovery between test preparation and reference preparation | up to 24 weeks
  Peak activity of FVIII (as Cmax) measured within 1 hour after the end of infusion.

SECONDARY OUTCOMES:
tmax | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on single dose in day 1 to day 4.
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of time to reach maximum plasma concentration
t1/2 | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on multiple dose in day 5 to day 8.
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of half-life
Mean time of residence (MRT) | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on single dose in day 1 to day 4.
  MRT is the average time that drug molecules stay in the body after a quick intravenous injection.
λz | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on single dose in day 1 to day 4.
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of terminal rate constant.
CL | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on single dose in day 1 to day 4.
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of apparent plasma clearance following intravenous injection.
Vz | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on single dose in day 1 to day 4.
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of apparent volume of distribution.
Area under the plasma concentration verus time curve (AUC) | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on multiple dose in day 5 to day 8.
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of area under the plasma concentration time curve from zero to infinity.
Peak plasma concentration (Cmax) | Hour 30min (pre-dose), 5min, 20min, 35min, 60min, 1.5 h, 2h, 3 h, 6 h, 9 h, 24 h, 36 h, 48 h post-dose on multiple dose in day 5 to day 8.
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of maximum plasma concentration.
Recombinant Coagulation Factor VIII multiple dose:tmax | On the 176th day after the prevention of medication
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of time to reach maximum plasma concentration.
Recombinant Coagulation Factor VIII multiple dose:t1/2 | On the 176th day after the prevention of medication
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of half-life.
Recombinant Coagulation Factor VIII multiple dose:λz | On the 176th day after the prevention of medication
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of terminal rate constant.
Recombinant Coagulation Factor VIII multiple dose:CL | On the 176th day after the prevention of medication
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of apparent plasma clearance following intravenous injection.
Recombinant Coagulation Factor VIII multiple dose:Vz | On the 176th day after the prevention of medication
  To characterize the pharmacokinetics of Recombinant Coagulation Factor VIII by assessment of apparent volume of distribution.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - AnHui Provincial Hospital, Hefei, Anhui
  - The First Hospital of LanZhou University, Lanzhou, Gansu
  - HeNan Cancer Provincial Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality